CLINICAL TRIAL: NCT00251966
Title: A Randomized Double-Blind Placebo-Controlled Study to Assess the Prevention of Low-Dose Acetylsalicylic Acid (ASA) Associated Gastroduodenal Lesions and Upper Gastrointestinal Symptoms in Patients Taking Esomeprazole 20 mg Once Daily for 26 Weeks.
Brief Title: ASTERIX: Low Dose ASA and Nexium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D9617C00011
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Gastroesophageal Reflux
Keywords: Prevention of gastroduodenal lesions; erosive oesophagitis; upper GI symptoms
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
The purpose of the study is to evaluate the effect of esomeprazole 20 mg od versus placebo for the prevention of gastric and/or duodenal ulcers in patients taking low-dose ASA.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of a condition (cardiovascular and/or cerebrovascular protection or other reasons) that requires daily intake of low-dose ASA, 75-325 mg, and is expected to continue for the duration of the study (daily is defined as at least 5 days per week).
* Age >= 60 years.
* No gastric and/or duodenal ulcer at the baseline endoscopy.
* H. pylori negative by serology test at screening.

Exclusion Criteria:

* Upper GI symptoms
* Erosive oesophagitis
* Malignancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960
Dates: Start 2004-05; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The primary variable is presence of gastric and/or duodenal ulcers at endoscopy over a 26-week period in patients taking low-dose ASA.

SECONDARY OUTCOMES:
LA classification for the oesophagus at endoscopy. Upper GI symptoms assessed by the investigator at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Science Director, MD, Study Director — AstraZeneca; Neville Yeomans, MD, Principal Investigator — Perth Medical School
Locations (94):
- Australia (9):
  - Research Site, Bondi Junction, New South Wales
  - Research Site, Bracken Ridge, Queensland
  - Research Site, Carina Heights, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Ashford, South Australia
  - Research Site, Wayville, South Australia
  - Research Site, Woodville, South Australia
  - Research Site, Ballarat, Victoria
  - Research Site, Malvern, Victoria
- Bulgaria (5):
  - Research Site, Burgas
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Canada (16):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Carbonear, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Thornhill, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Parkdale, Prince Edward Island
  - Research Site, Courcelette, Quebec
  - Research Site, Québec, Quebec
- Germany (30):
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, München, Bavaria
  - Research Site, Cottbus, Brandenburg
  - Research Site, Hamburg, Hamburg
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Hanover, Lower Saxony
  - Research Site, Rostock, Mecklenburg-Vorpommern
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Mainz, Rhineland-Palatinate
  - Research Site, Halle, Saxony-Anhalt
  - Research Site, Cologne
  - Research Site, Hamburg
  - Research Site, Herne
  - Research Site, Künzing
  - Research Site, Lienen
  - Research Site, Ludwigshafen
  - Research Site, Lüdenscheid
  - Research Site, Münster
  - Research Site, Oelde
  - Research Site, Paderborn
  - Research Site, Potsdam
  - Research Site, Ribnitz-Damgarten
  - Research Site, Rostock
  - Research Site, Siegen
  - Research Site, Wangen
  - Research Site, Wiesbaden
  - Research Site, Wolfenbüttel
  - Research Site, Wolmirstedt
  - Research Site, Zeven
- Greece (4):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Research Site, Hong Kong, Hong Kong
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Gy¿r
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Vác
- Italy (5):
  - Research Site, Bologna, BO
  - Research Site, Genova, GE
  - Research Site, Parma, PR
  - Research Site, Roma, Roma
  - Research Site, Napoli
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, Johannesurg
  - Research Site, Lyttelton Manor
  - Research Site, Parktown
  - Research Site, Tygerberg
- Spain (7):
  - Research Site, Santiago, A Coruña
  - Research Site, Santiago de Compostela, A Coruña
  - Research Site, Granada, Granada
  - Research Site, San Sebastián, Guipuzcoa
  - Research Site, Madrid, Madrid
  - Research Site, Murcia, Murcia
  - Research Site, Seville, Sevilla
- United Kingdom (4):
  - Research Site, Irvine, Ayrshire
  - Research Site, Glasgow, Scotland
  - Research Site, Cardiff, South Wales
  - Research Site, Edinburgh